CLINICAL TRIAL: NCT04907357
Title: rTMS for Stimulant Use Disorders (CTN-0108)
Brief Title: rTMS for Stimulant Use Disorders
Acronym: CTN-0108
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kathleen Brady, Distinguished University Professor, Department of Psychiatry and Behavioral Sciences, Medical University of South Carolina, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00107688; UG1DA013727 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Cocaine Use Disorder; Methamphetamine Abuse; Cocaine Dependence; Methamphetamine Dependence; Stimulant Use; Stimulant Abuse; Methamphetamine Use Disorder; Cocaine Abuse; Stimulant Use Disorder
Keywords: Stimulant; Cocaine; Methamphetamine; Repetitive Transcranial Magnetic Stimulation; rTMS
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is a double-blind, sham-controlled study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- rTMS (Active Comparator): Participants will receive up to 30 rTMS sessions within the 8-week treatment period.
  Interventions: Device: rTMS
- Sham (Placebo) (Sham Comparator): Participants will receive up to 30 sham rTMS sessions within the 8-week treatment period.
  Interventions: Device: Sham (Placebo)

INTERVENTIONS:
Device: rTMS — Each rTMS session will consist of 75 rTMS trains of 10 Hz for 4 seconds (40 pulses per train) with inter-train interval (ITI) of 11 seconds (a total of 3000 stimuli per session) over the left dorsolateral prefrontal cortex (DLPFC).
  Other Names: Repetitive Transcranial Magnetic Stimulation; TMS
  Arms: rTMS
Device: Sham (Placebo) — Each sham rTMS session will consist of 75 rTMS trains of 10 Hz for 4 seconds (40 pulses per train) with inter-train interval (ITI) of 11 seconds (a total of 3000 stimuli per session) over the left dorsolateral prefrontal cortex (DLPFC). In the placebo condition the magnetic field will be delivered in the opposite direction (away from the brain).
  Other Names: Sham Repetitive Transcranial Magnetic Stimulation
  Arms: Sham (Placebo)

SUMMARY:
The purpose of the study is to determine feasibility of repetitive transcranial magnetic stimulation (rTMS) for individuals with moderate to severe cocaine or methamphetamine use disorder (CUD/MUD). Potential participants will be age 18-65, and interested in cutting down or stopping use. Participants will be randomized to one of two groups; groups will receive rTMS or sham rTMS (placebo) over the course of an 8-week treatment period, and complete follow-up assessments at the end of treatment, 12, and 16 weeks post-randomization.

DETAILED DESCRIPTION:
The study will be a randomized, double-blind, sham-controlled trial comparing rTMS vs. placebo delivered over an 8-week treatment period. After assessment and inclusion into the study, participants will be randomized to receive up to 30 sessions of either rTMS or placebo treatments. The target minimum number of rTMS/placebo treatments is 20 treatments over 8 weeks. The secondary objective is to gather preliminary data on the efficacy of rTMS for individuals with moderate to severe CUD or MUD. Follow-up visits occur at end of treatment and at 12- and 16-weeks following randomization.

Other study procedures:

Actigraphy: To assess daily sleep quality during weeks 1-8, the ActiGraph wristband device will record, sleep latency, sleep duration, and intervals of waking during the sleep period.

Electroencephalography (EEG): EEG will be obtained after randomization and again at week 4, to explore the potential for EEG to be used as a biomarker of treatment response.

Cognitive-Behavioral Educational Intervention: Participants in both conditions (rTMS and placebo) will be encouraged to participate in a mobile app-based educational intervention based on principles of Cognitive Behavioral Therapy (CBT) for Substance Use Disorder (SUD).

Daily Assessments: Brief, electronic remote surveys will be administered to participants daily until week 16 follow-up time point and will assess use of primary substance of abuse, craving, ability to resist use, overall mood, and self-rated sleep quality.

Urine Drug Screens (UDS): UDS will be collected at screening, randomization, every treatment session, and at follow-up visits.

Urine pregnancy tests: Pregnancy testing for all female participants will be performed at screening, randomization, and monthly during the treatment period.

Physical exam: A physical exam will be performed at screening.

Questionnaires: A battery of study assessments will be completed to further inform findings regarding feasibility and effects of rTMS on individuals with stimulant use disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18-65, inclusive
* Have a diagnosis of moderate or severe Cocaine or Methamphetamine Use Disorder (CUD/MUD) over the past 12 months (as determined by DSM-5 diagnostic criteria).
* Have used cocaine or methamphetamine on at least 10 of the last 30 days (based on Timeline Follow-Back).
* Be interested in decreasing cocaine and/or methamphetamine use.
* If female, willing to use appropriate birth control method during the treatment phase of the study.
* Be able to understand the study procedures and provide written informed consent to participate in the study.
* If prescribed benzodiazepines or anticonvulsants, must be on a stable dose for at least 4 weeks prior to consent.

Exclusion Criteria:

* A Diagnostic and Statistical Manual (DSM-5) diagnosis of moderate or severe SUD of any substance other than cocaine or methamphetamine based on DSM-5.
* History of a serious medical disorder that, in the opinion of the Medical Clinician, would make it unsafe to participate in the study or may prevent collection of study data.
* Is currently engaged in formal SUD treatment.
* Documented history of unprovoked seizure (lifetime) or any seizure in the past 6 months.
* Documented history of brain lesion(s) and/or tumor(s).
* Metal implants or non-removable metal objects above the waist.
* Currently pregnant.
* Lifetime history of prior clinical treatment with TMS.
* Current or lifetime bipolar disorder.
* Current psychotic disorder or psychotic depression.
* Serious risk of homicide or suicide.
* Are a prisoner or in police custody at the time of eligibility screening.
* Previously randomized as a participant in the study.
* Planned admission to a residential treatment facility or other formal SUD treatment program.
* Unwilling or unable to follow study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen T Brady, MD PHD, Principal Investigator — Medical University of South Carolina; Madhukar Trivedi, MD, Principal Investigator — University of Texas South Western
Locations (4):
- United States (4):
  - Wake Forest, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The lead investigator will submit coded individual level data on Clinical Trials Network (CTN) study participants to the Data Management Center contracted by National Institute on Drug Abuse (NIDA) Center for CTN. These data may include but are not limited to: demographic information, date of birth, medical history, substance use history, psychiatric history, objective measures of substance use and psychiatric status, HIV status and genetic information. Data will be submitted without information that could readily identify the study participant (i.e. We will not share medical record numbers, social security numbers or participant names or phone numbers with the Data Management Center). De-identified data will be made publicly available per the CTN's policies
Supporting Information: Study Protocol
Time Frame: Data sets for this protocol will be available after (1) the primary paper has been accepted for publication, or (2) the data is locked for more than 18 months, whichever comes first.
Access Criteria: Prior to downloading any study data, the user will be prompted to complete a registration agreement for data use. Users will have to register a name and valid e-mail address in order to download data and to accept their responsibility for using data in accordance with the NIDA Data Share Agreement.
URL: https://datashare.nida.nih.gov

REFERENCES:
- [Derived] Atoui Z, Egan D, Jha MK, Hartwell K, Toll R, Sonne S, Brunner-Jackson B, Subramaniam G, McCauley JL, Trivedi M, Brady K. Repetitive transcranial magnetic stimulation for stimulant use disorders (STIMULUS): protocol for a multi-site, double-blind, randomized controlled trial. Addict Sci Clin Pract. 2025 May 8;20(1):40. doi: 10.1186/s13722-025-00567-w. PMID 40336040

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham (Placebo) | rTMS
Started | 63 | 66
Completed | 51 | 45
Not Completed | 12 | 21
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 9 | 18
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Unable to attend visits | 1 | 0
Not completed — Incarcerated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rTMS | Sham (Placebo) | Total
Number analyzed (Participants) | 66 | 63 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 62 | 127
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (9.38) | 46.8 (10.20) | 46.8 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 33
  Male | 46 | 50 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 19
  Not Hispanic or Latino | 55 | 55 | 110
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 26 | 28 | 54
  White | 32 | 30 | 62
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 66 | 63 | 129
Primary substance of use [Count of Participants; unit: Participants]
  Cocaine | 27 | 26 | 53
  Methamphetamine | 39 | 37 | 76
Major Depressive Episode [Count of Participants; unit: Participants] — Mini International Neuropsychiatric Interview (MINI) 7.0.2
  Participants
    Present | 5 | 4 | 9
    Absent | 61 | 59 | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Receive at Least 20 Sessions of rTMS/Sham Over the Treatment Period.
Description: Treatment session attendance and completion will be tracked over the course of the study, and this record will constitute the primary feasibility outcome.
Time Frame: From first treatment session (Week 1, first study visit) to end of treatment at 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | rTMS | Sham (Placebo)
Number analyzed (Participants) | 66 | 63
Participants
  Attended 20 or more rTMS/sham sessions | 29 | 40
  Attended fewer than 20 rTMS/sham sessions | 37 | 23

2. Secondary Outcome: Negative UDS From Weekly UDS
Description: A negative UDS for participants with cocaine as primary substance would be a UDS absent of cocaine; a negative UDS for participants with methamphetamine as primary substance would be a UDS absent of methamphetamine.
Time Frame: From first treatment week (Week 1) to end of treatment at 8 weeks
Measure: Number; unit: Urine drug screens
Units Other Than Participants: Urine drug screens
Arm/Group | rTMS | Sham (Placebo)
Number analyzed (Participants) | 66 | 63
Number analyzed (Urine drug screens) | 407 | 414
Urine drug screens
  Negative UDS | 38 | 30
  Positive UDS | 369 | 384

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Study specific SAEs are worsening depression, suicidal ideation, suicide attempt, suicide, hypomania/mania, seizure, and device malfunction resulting in injury.
  Study staff assesses for AEs and SAEs by asking the study participant, AEs and SAEs may also be spontaneously reported to study staff at any visit following consent. A suicide severity rating scale (CHRT) to assess both suicide intent and behavior was administered weekly during the treatment phase and at each follow-up visit.
Arm/Group | rTMS | Sham (Placebo)
All-Cause Mortality (participants affected / at risk) | 1/66 | 0/63
Serious Adverse Events (participants affected / at risk) | 5/66 | 2/63
Other Adverse Events (participants affected / at risk) | 45/66 | 29/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rTMS (N=66) | Sham (Placebo) (N=63)
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Cerebral vascular accident (Nervous system disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS (N=66) | Sham (Placebo) (N=63)
Headache (Nervous system disorders) | 7 (10) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (3) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (4)
Headache device related (Nervous system disorders) | 5 (11) | 6 (9)
Application site discomfort (General disorders) | 6 (7) | 2 (2)
Medical device site discomfort (General disorders) | 7 (7) | 5 (5)
Medical Device Site Pain (General disorders) | 19 (27) | 10 (12)
Blepharospasm device related (Eye disorders) | 4 (6) | 0 (0)
Muscle twitching device related (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (6)
Procedural Headache (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
Initial planned recruitment for the study was 160. An interim sample size re-estimation was completed and the targeted sample size was adjusted. A total of 129 individuals were randomized for participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT04907357/Prot_001.pdf
  • Statistical Analysis Plan (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT04907357/SAP_002.pdf
  • Informed Consent Form (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT04907357/ICF_000.pdf